CLINICAL TRIAL: NCT02845583
Title: Quantifying and Measuring the Economic Impact of Nursing Activities During the Hospital Stay of High Complexity Oncologic Care Patients
Brief Title: Nursing Activities for High Complexity Oncologic Care Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Amelia Palinuro, Phd Student, Catholic University of the Sacred Heart
Other Study IDs: FAG14
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Nursing; Diagnosis Related Group; Activity based costing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Retrospective cohort: 150 oncologic patients belonging to major complexity DRGs
- Perspective cohort: 150 oncologic patients belonging to major complexity DRGs

SUMMARY:
the study consists of an observational study aimed at quantifying the economic burden of the nursing activities on the overall cost of hospitalizations funded through DRG tariffs for Major complexity oncology patients.

DETAILED DESCRIPTION:
Study design

The methodological approach used to achieve the objective of this research is quantitative. A mixed study design is being adopted:

1. Retrospective study to determine the nature and volume of activity provided at nursing classes of patients whose admission is attributed to a specific DRG
2. Longitudinal prospective study to determine the variability of costs of nurses with regard to DRG refund, comparatively to distribution of patients for every single section (high, medium, low complexity).

Study population The sample has been chosen considering the prevalence of hospitalizations per year in medical oncology U.O.C. related to certain DRG and characterized by greater complexity of care, so as to provide a useful information base for study. For the retrospective study the survey will be conducted on a sample of 150 patients. Patients will be enrolled at high, medium and low complexity of care, hospitalized for chemotherapy and for biliary obstructive urinary tract and in the first half of 2016. It is estimated that the sample represents 30% of the total number of admissions made in 2016. A prospective longitudinal study will take into consideration a sample of 150 patients with the same characteristics considered for enrollment in the retrospective study.

The study will include patients who under go: CHT with a duration of hospital stay of 2-3 days (microcitomi and NHL), CHT with a length of hospital stay of 4-5 days (sarcomas), CHT with a length of hospital stay > 5 days or at high doses (testicle cancer, Ewing's sarcoma and bone sarcoma) and patients with higher complexity care.

Patients of 18 years of age or less will be excluded, as well as patients that were transferred to other units while inpatient, patients transferred in U.O.C. of Oncology after major surgery procedures in other departments, and admissions that are outliers.

The duration for the monitoring phase on the allocation and the distribution of patients among the different sections of hospital care intensity (Intensità di cure, IC) and care complexity (Complessità Assistenziale, CA), based on the results obtained by the Triage of corridor (TriCO), is estimated for 3 months up to a maximum of six months starting from March 2016. For the collection of data relating to the amount and types of activities provided in the first half of 2016 is estimated to have a maximum of 30 days and others 30 days for the detection the relative DRG reimbursed for hospitalizations considered.

Survey instruments

* Professional Assessment Instrument (PAI). It is a tool that documents nursing processes implemented in a computerized way using nursing language according to the North American Nursing Diagnosis Association International (NANDA-I).
* Hospital discharge card (Scheda di dimissione ospedaliera, SDO). It is a tool that contains information about each patient discharged, that are necessary for the attribution to DRG and for finding the rate payable for each episode of hospitalization
* Scheda di mobilità interna dei pazienti. It is a card that contains data of Tri-CO at the entrance of the patient and any variations of that index during hospitalization.

Interventions The study will be presented to the manager and coordinator of the U.O.C. Medical Oncology through a moment of training/information.

In order to collect data on the variation of Tri-CO during hospitalization, and consequently the different allocation to U.O.C. of Oncology of patients in sections of low, medium and high complexity of care, a point of contact (nurse) will be identified who will deal with the collection and retention of such information in the manner set out in the research protocol.

Outcome measures

The primary outcome expected by the survey is the quantification of the volume of nursing activities provided to patients and its cost. In addition, we expect to realize economic indicators which make it possible to ascertain:

* Cost weight of the nursing staff on the DRG rate reimbursed in relation to the complexity care of the patient;
* Cost weight of the nursing staff on the reimbursement for hospitalization in connection with the DRG of patient discharge.
* Gap between theoretical and actual cost of nurses in relation to the care delivered for a specific patient; Knowledge of actual costs for each distinct and specific episode of hospitalization would enhance its "uniqueness". An economic analysis of labor nursing costs for individual patient could provide input for the determination of the costs of all the professionals of the Foundation, contributing to the improvement of corporate strategic management for resource allocation.

Statistical analysis Statistical analyses will be performed using methods of descriptive statistics and inferential statistics appropriate to the sample size and study variables. Prospective longitudinal study will be used to determine the frequency distribution and the variance on the stay of the patients in each individual section of hospital in-patient treatment which is attributed to a specific DRG. Then a factorial analysis and regression techniques will be used to measure the type of bond that exists between the dependent variable Y (nursing) and independent variables X1, X2, X3 ... (DRG, age, days of hospitalization, complications, etc). Then the analysis will continue by studying which variables will affect the distribution of patients for IC and CA level and how it can change this assignment during a single in-patient episode, creating a variability in costs of services paid.

ELIGIBILITY:
Inclusion Criteria:

* CHT with a duration of hospital stay of 2-3 days (microcitomi and NHL),
* CHT with a length of hospital stay of 4-5 days (sarcomas),
* CHT with a length of hospital stay > 5 days (in case of high doses: testicle cancer, Ewing's sarcoma and bone sarcoma)
* Oncologic patients with higher complexity care.

Exclusion Criteria:

* Patients of 18 years of age or less
* Patients transferred to other units while inpatient
* Patients transferred in U.O.C. of Oncology after major surgery procedures in other departments
* Outlier admissions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample has been chosen considering the prevalence of hospitalizations per year in medical oncology U.O.C. related to certain DRG and characterized by greater complexity of care, so as to provide a useful information base for study. For the retrospective study the survey will be conducted on a sample of 150 patients. Patients will be enrolled at high, medium and low complexity of care, hospitalized for chemotherapy and for biliary obstructive urinary tract and in the first half of 2016.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Volume of Nursing Activity | Through study completion, based on the patients' discharge date. The first outcome assessments are expected in December 2016.
  Count of nusing activities performed to patients in different complexity groups

SECONDARY OUTCOMES:
Cost weight of the nursing staff on the DRG rate reimbursed in relation to the complexity care (Complessità Assistenziale, CA) of the patient. | Through study completion, based on the patients' discharge date. The first outcome assessments are expected in December 2016.
  Cost weight of the nursing staff on the DRG rate reimbursed in relation to the complexity care of the patient
Cost weight of the nursing staff on the reimbursement for hospitalization in connection with the DRG of patient discharge | Through study completion, based on the patients' discharge date. The first outcome assessments are expected in December 2016.
  Cost weight of the nursing staff on the reimbursement for hospitalization in connection with the DRG of patient discharge.
Mean difference between theoretical and actual cost of nurses in relation to the care delivered for a specific patient. | Through study completion, based on the patients' discharge date. The first outcome assessments are expected in December 2016.
  Difference between theoretical and actual cost of nurses in relation to the care delivered for a specific patient. The nursing time cost expressed in minutes results from the standard cost for each nursing hour worked by a nurse. The time in minutes of the performance is detected by the time indicated on standard nursing protocols considered for the study. The time in minutes of a benefit provided to specific types of patients considered comes from the average execution time of nursing care.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No